CLINICAL TRIAL: NCT06300853
Title: Understanding Adaptive Immune Response Elicited After COVID-19 Vaccination Boosters to Improve Vaccination Strategies in Vulnerable Groups.
Brief Title: Understanding Adaptive Immune Response After COVID-19 Vaccination Boosters to Improve Vaccination Strategies in Vulnerable Groups.
Acronym: COVaxFragile
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-07
Record Dates: First submitted 2024-03-06; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer patients (Other): Adult patients with a solid tumor diagnosis [I, II, III, IV stage,] and active anti-cancer treatment or treatment discontinued for less than 6 months, followed at IRCCS Sacro Cuore - Don Calabria, Negrar (Verona), Italy will be prospectively recruited at the moment of the future booster doses administration of SARS-CoV-2 vaccine.
  Interventions: Other: Analisys of cellular response and humoral response to SARS-CoV-2 vaccine booster doses
- Elderly subjects (Other): Subjects over 70 years of age who live in the nursing home in the social area at the IRCCS Sacro Cuore - Don Calabria Hospital will be prospectively recruited at the moment of the future booster doses administration of SARS-CoV-2 vaccine.
  Interventions: Other: Analisys of cellular response and humoral response to SARS-CoV-2 vaccine booster doses

INTERVENTIONS:
Other: Analisys of cellular response and humoral response to SARS-CoV-2 vaccine booster doses — Whole blood and serum samples will be longitudinally collected at the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1). Possible further time points will be collected within 2 years, based on the National recommended future vaccination regimens.
  Biological samples will be used for the following exams:
  * Cellular immunity characterization
    * T- and B-cells Immunophenotype.
    * Specific T-cell response.
    * In vitro specific B-cells characterization.
    * Antibody-dependent cellular cytotoxicity.
  * Humoral response characterization
    * Serology assays.
    * Avidity assay.
    * Neutralization assays with different SARS-CoV-2 variants.
    * Presence of specific or cross-reactive antibodies for common hCoV.
  * Genetic and epigenetic analysis

SUMMARY:
This is an experimental study without drug and device, non-profit, single-center.

The general objective of the project is to study how the adaptive immune response evolves against SARS-CoV-2 with repeated vaccination boosters and infections also in relation to the evolution of variations. This study will be relevant to frail populations who are the main targets of repeated vaccinations. Our project will benefit from the availability of a highly cohort characterized of vaccinated people, including cancer patients and elderly people, with prospective collection of samples for an in-depth evaluation of the evolution of the immune response with repeated exposure to doses of infection or vaccine. As part of the study, analyzes will be carried out on samples of patients enrolled in a manner prospective at the oncology departments of the IRCCS (Medical Oncology, Department of Radiotherapy advanced oncology and nuclear medicine) and elderly patients residing in retirement homes of the IRCCS. Patients will also be asked for consent to store any residual samples in the Tropica DITM Biobank.

ELIGIBILITY:
Cancer patients

Inclusion criteria:

* Age> 18 years.
* Solid tumor diagnosis [I, II, III, IV stage,].
* Vaccinated with anti-SARS-CoV-2 vaccine or/and having history of past SARS-CoV-2 infections.
* Signed informed consent.

Exclusion criteria

* Age < 18 years.
* Absence of signed informed consent.

Elderly subjects

Inclusion criteria:

* Age> 70 years.
* Vaccinated with anti-SARS-CoV-2 vaccine or/and having history of past SARS-CoV-2 infections.
* Signed informed consent.

Exclusion criteria

* Age < 70 years.
* Absence of signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Cellular response evaluation: flow cytometry profiles (proportions of cells) | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).
Cellular response evaluation: results of T and B cells stimulation with specific peptides (continuous variables, unity of measure: Optical Density OD) | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).
Cellular response evaluation: ADCC assay (continuous variables, unity of measure: Optical Density OD) | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).
Cellular response evaluation: anti-SARS-CoV-2 antibodies quantities (IgGs and IgM, BAU/ml) | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).
Cellular response evaluation: neutralization assays against different SARS-CoV-2 variants (continuous variables, unity of measure: TCID50/ml) | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).
Cellular response evaluation: avidity assays (continuous variables, unity of measure: BAU/ml). | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).
Humoral response evaluation: anti-SARS-CoV-2 antibodies quantities (IgGs and IgM, BAU/ml) | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).
  a) A b) Analysis results of , c) Analysis results of
Humoral response evaluation: neutralization assays against different SARS-CoV-2 variants (continuous variables, unity of measure: TCID50/ml) | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).
Humoral response evaluation: avidity assays (continuous variables, unity of measure: BAU/ml). | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).

SECONDARY OUTCOMES:
Neutralization assays against different human Coronavirus (hCoV). | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).
Whole genome sequencing analysis results | At the moment of the administration of the booster doses (T0) and three weeks after the booster doses (T1).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy